CLINICAL TRIAL: NCT03017287
Title: Safety and Efficacy of the GlucoMe APP in Patients With Uncontrolled Diabetes Treated With MDI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: GlucoMe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clin-002-00
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 1 or 2
Keywords: Glucose blood measurements, glucometer, BGM, Diabetes App
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GlucoMe App (Experimental): Self monitoring of glucose blood measurements using the GlucoMe glucose monitoring glucose device and App
  Interventions: Device: GlucoMe App

INTERVENTIONS:
Device: GlucoMe App — Assessment of the the GlucoMe App

SUMMARY:
The study will evaluate the safety and efficacy of computerized GlucoMe App in patients with uncontrolled diabetes treated with MDI.

DETAILED DESCRIPTION:
GlucoMe is an interactive system, which provides glucose management tools to both the patient and health care team (HCT). The system includes a decision support system to be used by the HCT aiming to aid clinical decision making with mathematical models. The system does not intend to replace clinical judgement and all recommendations are to be approved by the HCT.

Forty (40) diabetic patients on multiple daily insulin injection (MDI) with abnormal HbA1c and identified as potential end users of the device will be recruited to the study and screened according to the study inclusion and exclusion criteria. Patient's daily blood glucose will be measured and the GlucoMe App will give its recommendations for change in insulin dose, as well as recommendations for pre and post-meal carbohydrate and exercise. Patient's daily blood glucose levels will be followed by the HCT biweekly for 12 weeks and patients will be instructed to change their insulin doses according to the decision of the treating physician. At the end of the study, the HCT's recommendations for treatment adjustment will be compared to those of the system for both safety and efficacy. Study subjects and the HCT will be asked to complete a questionnaire regarding the GlucoMe system usability.

ELIGIBILITY:
Inclusion Criteria:

1. Both type 1 and type 2 diabetes
2. HbA1c 7-11%
3. Treated with MDI for at least 3 months
4. Ability to use the system at home, mobile phone

Exclusion Criteria:

1. Active CAD, CVA during last 6 months
2. Treatment with steroids or other glucose modifying drugs
3. Chronic infection/cancer/other severe disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Hypoglycemic and Hyperglycemic Events | At 12 weeks of the study
  Number and severity of hypoglycemic and severe hyperglycemic events
Correlation between GlucoMe and HCT recommendations | At 12 weeks of the study
  Correlation between GlucoMe and HCT recommendations for changing insulin dose and the treating physician/HCT advice.

SECONDARY OUTCOMES:
Target HbA1C/glucose achievement | At 12 weeks of the study
  Percent of patients that achieve HbA1C/glucose targets

CONTACTS AND LOCATIONS:
Locations (1):
- Diabitic Unit of the Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No